CLINICAL TRIAL: NCT02335892
Title: Patient Reported Outcomes With Fingolimod in Local Experience (PROFILE)
Brief Title: PROFILE - Evaluation of QoL and PRO Outcomes in Patients Taking Fingolimod
Acronym: PROFILE
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CFTY720DGB04
Record Dates: First submitted 2014-12-02; First posted 2015-01-12 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Multi centre, prospective, non interventional study in 200-240 UK relapsing remitting multiple sclerosis patients. Patients will complete questionnaires at baseline, 3, 6 and 12 months.

DETAILED DESCRIPTION:
Multi centre, prospective, non interventional study in 200-240 UK relapsing remitting multiple sclerosis patients assessing the change in QoL and PRO outcome measures from baseline to 12 months after starting fingolimod. Patients will complete 4 questionnaires at baseline (prior to first fingolimod dose), then repeat them at 3, 6 and 12 month intervals via post.

ELIGIBILITY:
Inclusion Criteria:

Patients prescribed Gilenya within the EU licence No previous exposure to Gilenya Patient's HCP considers patient able to complete study questionnaires Patient is between 18-55 years of age -

Exclusion Criteria:

There are no exclusion criteria for this study.

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with relapsing remitting multiple sclerosis starting treatment with fingolimod
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2014-11-11 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Changes from baseline after 12 months treatment with Gilenya as measured by the MSIS-29 (physical and psychological domains) | 12 months

SECONDARY OUTCOMES:
MSIS-29 and utility scores measured by EQ-5D-5L and any correlation between them | 12 months
Treatment Satisfaction Questionnaire for Medication (TSQM) and changes at 3 , 6 and 12mths after Gilenya treatment | 12 months
Morisky questionnaire and changes at 3 , 6 and 12 mths after treament with Gilenya | 12 months
Changes from baseline after 3 and 6 months treatment with Gilenya as measured by MSIS-29 | 12 months
Changes from Baseline after 3, 6 and 12 months of treatment with Gilenya as measured by EQ-5D-5L | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United Kingdom (11):
  - Novartis Investigative Site, Truro, Cornwall
  - Novartis Investigative Site, Swansea, England
  - Novartis Investigative Site, Romford, Essex
  - Novartis Investigative Site, Basingstoke, Hampshire
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Nottingham